CLINICAL TRIAL: NCT05836064
Title: GastroBot: a New Artificial Intelligence-developed Software Bot to Improve Bowel Preparation and Colonoscopy Quality
Brief Title: GastroBot: Artificial Intelligence Applied to Bowel Preparation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Institute of Gastroenterology and Advance Endoscopy (Other)
Responsible Party: Principal Investigator, Manuel Valero, Medical director, Institute of Gastroenterology and Advance Endoscopy
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Diagnostic
Other Study IDs: IGEA01-2023
Record Dates: First submitted 2023-04-18; First posted 2023-05-01 (Actual); Last update posted 2023-11-24 (Actual); Status verified 2023-11

CONDITIONS: Colonic Polyp; Colonic Neoplasms; Colonic Disease; Colonic Adenoma
Keywords: bowel preparation; colonoscopy quality
MeSH Terms: conditions — Colonic Polyps; Colonic Neoplasms; Colonic Diseases

STUDY DESIGN:
Intervention Model Description: The following is a cross-section simple-blind and single-center controlled randomized trial. Two groups will be established: the GastroBot-assisted bowel preparation (GB-group) and the conventional-assisted bowel preparation (C-group) group. Patients from both study groups will receive the same type of preparation with polyethylene glycol in split dose, establishing the intake time according to three-time segments (8-11 am, 11-2 pm, 2-4 pm).
Who Masked: Investigator, Outcomes Assessor
Masking Description: A clinical coordinator will be responsible for patients' randomization. The endoscopist will perform the endoscopy by assessing primary and secondary endpoints, blinded to the patient's study group.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- GastroBot-assisted bowel preparation group (GB-group) (Experimental): Adult patients with no surgical high-risk comorbidities and colonoscopy indications for screening, surveillance, or diagnosis who are undergoing a colonoscopy. GastroBot assisted with the polyethylene glycol bowel preparation: patients will receive the instructions through the WhatsApp application, being guided by the software bot with multiple and personalized alternative instructions according to results.
  Interventions: Device: GastroBot
- Conventional-assisted bowel preparation group (C-group). (Experimental): Adult patients with no surgical high-risk comorbidities and colonoscopy indications for screening, surveillance, or diagnosis who are undergoing a colonoscopy. The patients received bowel polyethylene glycol bowel preparation instructions in writing without prior personalized advice.
  Interventions: Other: Conventional explanation

INTERVENTIONS:
Device: GastroBot — An artificial intelligence-developed and WhatsApp-based software bot. It will send the instructions to the patient through the WhatsApp application, guided by the software bot with multiple and personalized alternative instructions according to results.
  Arms: GastroBot-assisted bowel preparation group (GB-group)
Other: Conventional explanation — Patients will receive in writing detailed explanation about bowel preparation with polyethylene glycol
  Arms: Conventional-assisted bowel preparation group (C-group).

SUMMARY:
It is estimated that about 20% of colonoscopies have inadequate preparation. (5) This is associated with lengthy procedures and less detection of adenomas, reduces the screening intervals, and increases the costs and risks of complications. Several strategies have been proposed to improve the quality of bowel preparation. Mobile healthcare Apps have been developed to increase adherence to bowel preparation agents, improving the quality of bowel preparation. However, adherence to mobile healthcare Apps is also a quality criterion and a pending problem to solve with this new technology.

GastroBot is a new technology based on artificial intelligence that allows, through a software bot, to carry out a personalized follow-up of the patient's bowel cleansing, advising the patient to overcome contingencies that arise with the preparation, which in other circumstances could lead to the failure of it. The primary aim of this study is to determine the improvement in bowel preparation after GastroBot assistance compared with the traditional explanation. As a secondary aim, this study also pursues to determine adenoma and polyp detection rates (ADR and PDR, respectively), bowel preparation agents' tolerance, and GastroBot functionality.

DETAILED DESCRIPTION:
Background Colorectal cancer (CRC) is the third most frequent tumor, the most frequent gastrointestinal tumor, and the second cause of cancer-related death. (1) In more than 80-90% of cases, CRC has a precursor lesion, an adenomatous polyp or adenoma, slowly progressing towards CRC. Colonoscopy is considered the gold standard in its prevention since it allows the detection and treatment of its initial form. (2) Considering this, several colonoscopy quality indicators have been described, such as cecal intubation rate, withdrawal time, and adenoma/polyp detection rate (ADR); the last is the most important indicator correlating with CRC risk. (3)

Therefore, focusing on improving the ADR is mandatory to reduce the incidence of CRC. Many techniques have been described for this purpose, like improving endoscopists' education and training, split-dosing bowel preparations, withdrawal time >9 minutes and right colon second view, high-definition white light endoscopy, Endocuff vision, G-EYE scope or Artificial Intelligence. (2, 4) However, all these techniques have in common the need for optimal visualization of the intestinal mucosa, which depends on bowel cleansing. (3,4)

Problem It is estimated that about 20% of colonoscopies have inadequate preparation. (5) This is associated with lengthy procedures and less detection of adenomas, reduces the screening intervals, and increases the costs and risks of complications. This causes frustration for the patient and physician with medico-legal conflicts. (6) The ideal cleansing method must be safe, well-tolerated, and effective. However, none of the current options fulfills these characteristics. The main cause of inappropriate cleansing (80% of cases) is a failure to adequately follow preparation instructions and mostly because of intolerance to the oral solution. (7,8)

Several strategies have been proposed to improve the quality of bowel preparation. As in other fields, mobile healthcare Apps have been developed to increase adherence to bowel preparation agents, improving quality bowel preparation. However, adherence to mobile healthcare Apps is also a quality criterion and a pending problem to solve with this new technology. Also, as with any mobile App, mobile healthcare Apps must be compatible with specific devices. GastroBot is a new technology based on artificial intelligence that allows, through a software bot, to carry out a personalized follow-up of the patient's bowel cleansing, advising the patient to overcome contingencies that arise with the preparation, which in other circumstances could lead to the failure of it.

Aim The primary aim of this study is to determine the improvement in bowel preparation after GastroBot assistance compared with the traditional explanation. As a secondary aim, this study also pursues to determine adenoma and polyp detection rates (ADR and PDR, respectively), bowel preparation agents' tolerance, and GastroBot functionality.

MATERIALS AND METHODS

Study design Study type. The following is a cross-section simple-blind and single-center controlled randomized trial. Two groups will be established: the GastroBot-assisted bowel preparation (GB-group) and the conventional-assisted bowel preparation (C-group) group.

Setting. It will be performed in consecutive patients with bowel preparation agents indication before undergoing a colonoscopy with cecal intubation at the Instituto de Gastroenterología y Endoscopía de Avanzada (IGEA), Hospital de la Asociación Médica (HAM) "Dr. Felipe Glasman" Bahía Blanca, Buenos Aires province, Argentina. The study protocol and consent form have been approved by the Institutional Review Board (IRB) and will be conducted according to the declaration of Helsinki. Patients will sign an informed consent.

Intervention A clinical coordinator will be responsible for patients' randomization. Patients from both study groups will receive the same type of preparation with polyethylene glycol in split dose, establishing the intake time according to three-time segments (8-11 am, 11-2 pm, 2-4 pm). The C-group will receive the instructions in writing without prior personalized advice. The GB group will receive the instructions through the WhatsApp application, guided by the software bot with multiple and personalized alternative instructions according to results. The endoscopist will perform the endoscopy by assessing primary and secondary endpoints, blinded to the patient's study group.

Sample size Considering the proportion of insufficient BBPS (<6) among the App-group (7.7%) vs. controls (16.9%) described by Walter B et al. (2021), a sample size of 194 cases per study group was estimated to determine a two-sided difference on BBPS between GB-group vs. C-group with an 80% statistical power.

Statistical analysis Baseline characteristics will be compared between the case and control group using Chi-square o Fisher test for categorical variables and Mann-Whitney U or Student's t-test for continuous variables. A P value of less than 0.05 will be considered statistically significant. All the statistical analysis will be performed using the latest version of the statistical program R (R Foundation for Statistical Computing; Vienna, Austria).

Limitations The protocol will be performed in only one center and by six endoscopists. It is a simple blind study. The patients will know they are using (or not) a novel instrument to increase bowel preparation quality.

ELIGIBILITY:
Inclusion Criteria:

* Age under 18 and over 80 years old.
* Who agrees to participate in the study and can understand and provide written informed consent.
* Any colonoscopy indication: colorectal neoplasia screening, surveillance of colon pre-existing diseases, or diagnostic approach in symptomatic patients.
* Smartphone owners (any device) and WhatsApp users, independence of local or international mobile phone provider.

Exclusion Criteria:

* Scheduled colonoscopies with any therapeutic approach will be categorically excluded if it does not have a cecal intubation indication.
* Patients with difficulty understanding instructions for bowel preparation or not being able to use WhatsApp.
* History of diabetes mellitus with insulin therapy, heart disease, kidney, liver, or severe metabolic disorder.
* Phenprocoumon therapy or severe uncontrolled coagulopathy
* Pregnancy and lactation
* Prior history of colon resection, ileostomy, or colostomy

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 388 (Estimated)
Dates: Start 2024-01-01 (Estimated); Primary Completion 2024-12-01 (Estimated); Study Completion 2025-04-28 (Estimated)

PRIMARY OUTCOMES:
Colonoscopy cleansing in terms of Boston bowel preparation score (BBPS) | 1 hour
  Visual assessment of colonoscopy cleansing per colonic part (left, transverse, right), based on BBPS scale.
Re-scheduled colonoscopy | 1 hour
  If bowel preparation was enough unsatisfactory to re-scheduled colonoscopy.

SECONDARY OUTCOMES:
Colonoscopy entrance time | 1 hour
  Time since colonoscopy beginning to cecal visualization.
Adenoma and polyp detection | 1 hour
  Visualization of any adenoma or polyp during colonoscopy
Bowel preparation agent's tolerance | 1 hour
  Any adverse event related to polyethylene glycol intake
GastroBot functionality | 1 hour
  Patient's qualification of his/her interaction with GastroBot, in accordance with the Mobile App Rating Survey scale (MARS). Due that GastroBot is not a proper App, only MARS functionality questions will be given to the patient, an only patients from the GB group.

CONTACTS AND LOCATIONS:
Overall Officials: Manuel Valero, MD, Principal Investigator — Instituto de Gastroenterología y Endoscopía de Avanzada (IGEA)
Locations (1):
- Institute of Gastroenterology and Advanced Endoscopy (IGEA), Bahía Blanca, Buenos Aires, Argentina

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gubbiotti A, Spadaccini M, Badalamenti M, Hassan C, Repici A. Key factors for improving adenoma detection rate. Expert Rev Gastroenterol Hepatol. 2022 Sep;16(9):819-833. doi: 10.1080/17474124.2022.2128761. Epub 2022 Oct 14. PMID 36151898
- [Background] Rex DK, Schoenfeld PS, Cohen J, Pike IM, Adler DG, Fennerty MB, Lieb JG 2nd, Park WG, Rizk MK, Sawhney MS, Shaheen NJ, Wani S, Weinberg DS. Quality indicators for colonoscopy. Gastrointest Endosc. 2015 Jan;81(1):31-53. doi: 10.1016/j.gie.2014.07.058. Epub 2014 Dec 2. No abstract available. PMID 25480100
- [Background] Hassan C, Spadaccini M, Iannone A, Maselli R, Jovani M, Chandrasekar VT, Antonelli G, Yu H, Areia M, Dinis-Ribeiro M, Bhandari P, Sharma P, Rex DK, Rosch T, Wallace M, Repici A. Performance of artificial intelligence in colonoscopy for adenoma and polyp detection: a systematic review and meta-analysis. Gastrointest Endosc. 2021 Jan;93(1):77-85.e6. doi: 10.1016/j.gie.2020.06.059. Epub 2020 Jun 26. PMID 32598963
- [Background] Ness RM, Manam R, Hoen H, Chalasani N. Predictors of inadequate bowel preparation for colonoscopy. Am J Gastroenterol. 2001 Jun;96(6):1797-802. doi: 10.1111/j.1572-0241.2001.03874.x. PMID 11419832
- [Background] Aganiants EK. [Changes in the impulse activity of cerebral cortex neurons upon inhalation of ether in different concentrations]. Biull Eksp Biol Med. 1968 Sep;66(9):45-8. No abstract available. Russian. PMID 5758907
- [Background] Jansen SV, Goedhard JG, Winkens B, van Deursen CT. Preparation before colonoscopy: a randomized controlled trial comparing different regimes. Eur J Gastroenterol Hepatol. 2011 Oct;23(10):897-902. doi: 10.1097/MEG.0b013e32834a3444. PMID 21900786
- [Background] Juluri R, Eckert G, Imperiale TF. Polyethylene glycol vs. sodium phosphate for bowel preparation: a treatment arm meta-analysis of randomized controlled trials. BMC Gastroenterol. 2011 Apr 14;11:38. doi: 10.1186/1471-230X-11-38. PMID 21492418
- [Background] Hassan C, East J, Radaelli F, Spada C, Benamouzig R, Bisschops R, Bretthauer M, Dekker E, Dinis-Ribeiro M, Ferlitsch M, Fuccio L, Awadie H, Gralnek I, Jover R, Kaminski MF, Pellise M, Triantafyllou K, Vanella G, Mangas-Sanjuan C, Frazzoni L, Van Hooft JE, Dumonceau JM. Bowel preparation for colonoscopy: European Society of Gastrointestinal Endoscopy (ESGE) Guideline - Update 2019. Endoscopy. 2019 Aug;51(8):775-794. doi: 10.1055/a-0959-0505. Epub 2019 Jul 11. PMID 31295746
- [Background] Walter B, Frank R, Ludwig L, Dikopoulos N, Mayr M, Neu B, Mayer B, Hann A, Meier B, Caca K, Seufferlein T, Meining A. Smartphone Application to Reinforce Education Increases High-Quality Preparation for Colorectal Cancer Screening Colonoscopies in a Randomized Trial. Clin Gastroenterol Hepatol. 2021 Feb;19(2):331-338.e5. doi: 10.1016/j.cgh.2020.03.051. Epub 2020 Mar 30. PMID 32240835